CLINICAL TRIAL: NCT05520372
Title: Evaluating Safety and Quality of Life of Cancer Patients Treated by Autologous Immune Enhancement Therapy (AIET) in Vinmec International Hospitals
Brief Title: Autologous Immune Enhancement Therapy (AIET) for Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIET_2022
Record Dates: First submitted 2022-08-23; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Patients With Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- autologous immune enhancement therapy (AIET) for treating cancer (Experimental): A total of 60 cancer patients received one to seven sittings of natural killer (NK) cells and cytotoxic T lymphocytes (CTLs) infusions.
  Interventions: Combination Product: Autologous immune enhancement therapy (AIET) for cancer patients

INTERVENTIONS:
Combination Product: Autologous immune enhancement therapy (AIET) for cancer patients — Autologous NK cell and CD8 T cell therapy for cancer patients

SUMMARY:
This is a retrospective study that included 60 cancer patients who underwent autologous NK cell and CD8 T cell therapy between January 2016 and December 2021

DETAILED DESCRIPTION:
The dysfunction and reduced proliferation of peripheral immune cells including CD8 T and NK cells have been observed in both aging and cancer patients, thereby challenging the immune cell therapy in these subjects. Therefore, we evaluated the growth of these lymphocytes in elderly patients with several types of cancer and the correlation of peripheral blood (PB) indexes to the expansions. This is a retrospective study that included 60 cancer patients who underwent autologous NK cell and CD8 T cell therapy between January 2016 and December 2021. By optimizing the antiviral and tumor surveillance ability of both NK cells and CTLs through serial steps from isolation and expansion, followed by re-infusion of these activated cells back to the patient body, AIET has become a promising, cutting-edge method in detecting and eliminating cancer cells. The study aimed to evaluate the safety and effectiveness of 60 cancer patientsreceiving AIET.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 75
* Patients have been diagnosed with cancer.
* Patients signed the written informed consent form.

Exclusion Criteria:

* Severe health conditions such as serious infection, autoimmune diseases, or using any anti-rejection drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events and serious adverse events (AEs or SAEs) | up to the 36-month period following treatment
  the number of AEs or SAEs during and after Autologous Immune Enhancement Therapy (AIET)

SECONDARY OUTCOMES:
Changes in health-related quality of life of patients | up to the 36-month period following treatment
  Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Version 3.0
Survival time of patients in this study | up to the 36-month period following treatment
  Survival time was defined as from the date of diagnosis until death or the end of this study
Changes in Symptoms of patients using MD Anderson Symptoms Inventory Gastrointestinal Cancer Module (MDASI ) | up to the 36-month period following treatment
  MDASI contains a 24-item questionnaire. MDASI-GI symptom items are assessed on a numeric scale ranging from 0 or "not present" to 10 or "as bad as you can imagine". The MDASI is a concise, internally stable, and sensitive tool for measuring multiple-symptom severity and symptom interference with function in patients with cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Liem Nguyen Thanh, PhD, Principal Investigator — Vinmec Research Institute of Stem Cell and Gene Technology
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No